CLINICAL TRIAL: NCT01470508
Title: Engaging Latino Families in Eating Disorders Treatment
Acronym: PAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mae Lynn Reyes-Rodriguez, PhD (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); National Institute of Mental Health (NIMH) (NIH); El Futuro (Other)
Responsible Party: Sponsor-Investigator, Mae Lynn Reyes-Rodriguez, PhD, Clinical Assistant Professor in Psychiatry, University of North Carolina, Chapel Hill
Organization: University of North Carolina, Chapel Hill (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-0773; IRB# 10-0773 (Other: University of North Carolina Institutional Review Board); K-23-MH087954-01A1 (Other Grant/Funding Number: NIMH)
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Bulimia Nervosa; Binge Eating Disorder; Eating Disorder Not Otherwise Specified
Keywords: Bulimia; Binge-Eating Disorder; Eating Disorders
MeSH Terms: conditions — Bulimia Nervosa; Binge-Eating Disorder; Bulimia; Feeding and Eating Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family Enhancement (Experimental): PAS is a 27-week program consisting of 25 sessions, 50 minutes in length, between an individual and a therapist. During six (6) family sessions, a family member will accompany the individual to therapy and will take an active role during the session. In this program, individuals and their family members will learn about ways to communicate about their relationship in the context of experiencing an eating disorder. PAS focuses on family-specific skills such as communication skills and problem solving skills while also incorporating eating disorders psychoeducation.
  Interventions: Behavioral: Cognitive Behavioral Therapy with Family Enhancement
- Cognitive Behavioral Therapy (Active Comparator): Individuals meet their therapist once a week for 25 sessions, 50 minutes in length, for a period of 27 weeks for therapy.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Individuals meet with a therapist once a week for 25 sessions, 50 minutes in length, for a period of 27 weeks for therapy. Cognitive Behavioral Therapy is manualized and is the standard form of care at the UNC Eating Disorders Program.
  Other Names: Eating disorder treatment as usual
  Arms: Cognitive Behavioral Therapy
Behavioral: Cognitive Behavioral Therapy with Family Enhancement — Individuals will meet with a therapist once a week for 25 sessions, 50 minutes in length, for a period of 27 weeks for therapy. Cognitive Behavioral Therapy with Family Enhancement is manualized and will involve the participation of family members during six (6) weeks of treatment.
  Other Names: PAS
  Arms: Family Enhancement

SUMMARY:
Promoviendo Alimentacion Saludable (PAS)"Promoting Healthy Eating" is a research project funded by the National Institute of Mental Health. The purpose of this study is to develop and test a treatment for eating disorders in Latina adults that is appropriate for their age and includes culturally appropriate family intervention.

DETAILED DESCRIPTION:
Research on culturally sensitive assessment and treatment of eating disorders among Latinos is scarce. This study is comparing individual Cognitive Behavioral Therapy (CBT) versus CBT with a family adjunctive intervention for eating disorders in Latina adults. All treatment will be conducted by trained professionals from either the UNC Eating Disorders Program (in Chapel Hill) or from El Futuro, Inc. (in Carrboro or Durham, NC) who have been trained in the treatment of eating disorders.

Participants will participate in 25, 50 minute-long, face-to-face CBT sessions over 27 weeks. Participants will be randomly placed in one of two groups: CBT or CBT with family enhancement. Those participants who are randomly placed into the CBT group will participate in 25 individual therapy sessions, 3 sessions with a dietitian, and psychiatry and/or medical assessments as needed. Those participants who have been randomly placed into the CBT with family enhancement group will participate in 19 individual therapy sessions, 6 family therapy sessions, 3 sessions with a dietitian, and psychiatry and/or medical assessments as needed. All participants will also be expected to participate in baseline, week 6 (mid-treatment), end of treatment, and 3-month follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV criteria for BN, BED, EDNOS (sub-threshold BN)
* Latina
* If taking antidepressant medication, stable dose for at least 3 months prior
* Willingness to ask a family member or significant other to participate AND agreement of family member to participate

Exclusion Criteria:

* Any major medical condition that would interfere with treatment or require alternative treatment
* Alcohol or drug dependence in the last three months
* Current significant suicidal ideation
* Developmental disability that would impair the ability of the participant to benefit from psychotherapy effectively
* Psychosis, including schizophrenia, or bipolar I disorder
* Pregnancy
* Body mass index below 17.5 kg/m^2
* If taking antidepressant medication, doses are not stable; individuals taking any medications that can significantly affect appetite or weight.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Eating Disorder Examination (EDE) Scores at End of Treatment | Baseline, End of Treatment
  End of Treatment will be measured by the completion of the twenty-five (25) scheduled therapy session, regardless of treatment group.

SECONDARY OUTCOMES:
Change from Baseline in Beck Depression Inventory-Revised (BDI-R) score at Week 6 of Treatment | Baseline, Week 6
Change from Baseline in Beck Depression Inventory-Revised (BDI-R) score at End of Treatment | Baseline, End of Treatment
  End of Treatment will be measured by the completion of the twenty-five (25) scheduled therapy session, regardless of treatment group.
Change from Baseline in Beck Depression Inventory-Revised (BDI-R) score at 3 Month Follow-up | Baseline, 3 Month Follow-up
Change from Baseline in the Symptom Checklist-36 (SCL-36) score at Week 6 of Treatment | Baseline, Week 6 of Treatment
Change from Baseline in Symptom Checklist-36 (SCL-36) score at End of Treatment | Baseline, End of Treatment
  End of Treatment will be measured by the completion of the twenty-five (25) scheduled therapy session, regardless of treatment group.
Change from Baseline in Symptom Checklist-36 (SCL-36) score at 3 Month Follow-up | Baseline, 3 Month Follow-up
Change from Baseline in Family Support Questionnaire score at End of Treatment | Baseline, End of Treatment
  End of Treatment will be measured by the completion of the twenty-five (25) scheduled therapy session, regardless of treatment group.
Change from Baseline in Family Support Questionnaire score at 3 Month Follow-up | Baseline, 3 Month Followup
Change from Baseline in Family Cohesion (FC) score at End of Treatment | Baseline, End of Treatment
  End of Treatment will be measured by the completion of the twenty-five (25) scheduled therapy session, regardless of treatment group.
Change from Baseline in Family Cohesion (FC) score at 3 Month Follow-up | Baseline, 3 Month Follow-up
Change from Baseline in Family Burden Interview Scale (FBIS) score at End of Treatment | Baseline, End of Treatment
  End of Treatment will be measured by the completion of the twenty-five (25) scheduled therapy session, regardless of treatment group.
Change from Baseline in Family Burden Interview Scale (FBIS) score at 3 Month Follow-up | Baseline, 3 Month Follow-up
Change from Baseline in Family Score (FS) at End of Treatment | Baseline, End of Treatment
Change from Baseline in Family Score (FS) at 3 Month Follow-up | Baseline, 3 Month Follow-up
Treatment Adherence as of End of Treatment | Baseline, End of Treatment
  Treatment Adherence will be measured positively if a participant has completed at least 80% of treatment (20 sessions or more) or negatively if less than 80% of treatment (19 sessions or less) has been completed.
Change from Baseline in Eating Disorder Examination Questionnaire (EDE-Q) score at Week 6 of Treatment | Baseline, Week 6
Change from Baseline in Eating Disorder Examination Questionnaire (EDE-Q) score at End of Treatment | Baseline, End of Treatment
  End of Treatment will be measured by the completion of the twenty-five (25) scheduled therapy session, regardless of treatment group.
Change from Baseline in Eating Disorder Examination Questionnaire (EDE-Q) score at 3 Month Follow-up | Baseline, 3 Month Follow-up

OTHER OUTCOMES:
M-FED Questionnaire | 3 Month Follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Mae Lynn Reyes-Rodriguez, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - University of North Carolina, Chapel Hill, North Carolina
  - UNC Center of Excellence for Eating Disorders, Chapel Hill, North Carolina